CLINICAL TRIAL: NCT01150916
Title: B-type Natriuretic Peptide in the Diagnosis of Heart Failure Related Ascites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Alberto Queiroz Farias, M.D. P.h.D., University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: CapPesq0074/10
Record Dates: First submitted 2010-06-23; First posted 2010-06-28 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Heart Failure; Liver Cirrhosis; Ascites; Carcinomatosis
Keywords: natriuretic peptide; heart failure; ascites; liver cirrhosis
MeSH Terms: conditions — Heart Failure; Liver Cirrhosis; Ascites; Carcinoma

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- Heart failure (Active Comparator): Patients must fulfill Framingham and/or Boston criteria for heart failure and have systolic or diastolic disfunction in rest echocardiography.
  Interventions: Procedure: BNP, SAAG, ascites total protein, echocardiography
- Liver Cirrhosis (Active Comparator): Patients must have a biopsy proven diagnosis of liver cirrhosis or the diagnosis established on clinical basis in cases of known etiology of liver disease, peripheral signs of chronic liver disease, esophageal varices at endoscopy and an imaging method with evidence of cirrhosis.
  Interventions: Procedure: BNP, SAAG, ascites total protein, echocardiography
- Other causes of ascites (Active Comparator): Patients must fulfill stringent diagnostic criteria for the cause of ascites, by clinical criteria, laboratory and imaging tests and histology when appropriate.
  Interventions: Procedure: BNP, SAAG, ascites total protein, echocardiography
- Concurrent heart failure and cirrhosis (Active Comparator): Patients must fulfill the aforementioned criteria for both conditions.
  Interventions: Procedure: BNP, SAAG, ascites total protein, echocardiography

INTERVENTIONS:
Procedure: BNP, SAAG, ascites total protein, echocardiography — diagnostic tests
  Other Names: BNP kit ADVIA Centaur BNP Siemens Inc, San Diego, CA, USA

SUMMARY:
The serum albumin ascites gradient (SAAG) is a recommended tool for ascites diagnosis since values ≥1.1 g/dl are found in nearly 97% of patients with portal hypertension. However, it mislabels chronic liver disease and heart failure as the cause of ascites. Because type-B Natriuretic Peptide (BNP) is increased in several body fluids of patients with both systolic and diastolic dysfunction, it was found to be a useful marker for diagnosing heart failure and pleural effusion due to heart failure. Nevertheless, to date, the performance of BNP testing for assessing the etiology of ascites has not been examined. The current prospective study is aimed at comparing the following strategies for diagnosing heart failure as the cause of ascites: 1) SAAG plus total protein concentration in ascitic fluid (gold standard); 2) SAAG plus BNP concentration in ascitic fluid; 3) SAAG plus BNP concentration in serum; 4) serum BNP concentrations.

SAAG, ascitic fluid protein concentration, serum and ascites type-B Natriuretic Peptide and echocardiography will be performed in all patients. The final diagnosis of the cause of ascites will be adjudicated by independent physicians, blinded for the results of ascitic fluid biochemistry and BNP. Patients will be divided into four groups: Heart failure, Liver cirrhosis, concurrent heart failure and liver cirrhosis (mixed) and other causes of ascites.

DETAILED DESCRIPTION:
Diagnostic criteria for the cause of ascites - two independent cardiologists and two hepatologists will interview and examine the enrolled patients and review the clinical records, laboratory and imaging findings to adjudicate the correct final cause of the ascites. They will have access to all exams that patients undergo, including results of biopsies, laboratory tests, chest radiography, Doppler ultrasound, computerized tomography, magnetic resonance imaging, echocardiography and cardiac catheterism. Liver cirrhosis diagnosis will be biopsy proven or established on clinical basis in patients with known etiology of liver disease, peripheral signs of chronic liver disease, esophageal varices at endoscopy and a compatible imaging method. Heart failure will be diagnosed in patients fulfilling Framingham and/or Boston criteria and by rest echocardiography. Other causes of ascites will be diagnosed by appropriate laboratory and imaging tests and by histology when appropriate.

SAAG, ascitic fluid protein concentration and type-B Natriuretic Peptide - will be assessed in all patients. BNP measurements will be carried out according to the instructions of the manufacturer in fresh samples (ADVIA Centaur BNP Siemens Inc, San Diego, CA, USA). This assay is a fully automated two-site sandwich immunoassay based on chemiluminescent technology, standardized with synthetic purified protein preparation of human BNP (aminoacid 77 to 108), for quantitative BNP within the range of <2.0 to 5,000 pg/ml. The BNP assay is reliable in presence of increased values of several biochemical parameters usually found in patients with decompensated cirrhosis. No interference in measurement has been reported from urea up to 200 mg/dL, creatinine up to 2.5 mg/dL, unconjugated bilirubin up to 25 mg/dL, conjugated bilirubin up to 25 mg/dL, triglycerides up to 800 mg/dL, cholesterol up to 1000 mg/dL and from commonly used pharmaceutical drugs. For testing in whole blood, a 4 ml sample will be collected in an EDTA containing tube. A 10 ml of ascitic fluid will be collected at the same time by paracentesis before infusion of albumin or volume overload. Laboratory staff will be unaware of both the clinical diagnosis and routine laboratory results.

Echocardiography - will performed at rest in all patients for assessing the following parameters: ejection fraction, left atrium diameter, systolic and diastolic left ventricle diameter and diastolic dysfunction.

Base-line demographical,past medical history and laboratory test results of all patients will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years old.
* must have signed the written informed consent.
* ascites of any etiology on clinical and laboratory imaging.
* fulfil stringent diagnostic criteria for the cause of the ascites.

Exclusion Criteria:

* contra-indication for paracentesis (hemodynamic instability, shock, active variceal bleeding etc).
* sepsis.
* fulminant liver failure.
* pregnancy.
* history of recent transfusion of blood components and/or derivates or volume expansion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2010-06; Primary Completion 2011-11 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
diagnostic accuracy of BNP for the diagnosis of ascites due to heart failure | 6 months
  * ROC curves of different strategies with and without BNP levels for diagnosing heart failure as the cause of ascites.
  * Sensitivity, specificity, accuracy, predictive values, likelihood ratios.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Q. Farias, MD, PhD, Principal Investigator — University of Sao Paulo School of Medicine
Locations (2):
- Brazil (2):
  - Federal University of Espirito Santo, Vitória, Espírito Santo
  - Hospital das Clinicas. University of São Paulo, São Paulo, São Paulo

REFERENCES:
- [Derived] Farias AQ, Silvestre OM, Garcia-Tsao G, da Costa Seguro LF, de Campos Mazo DF, Bacal F, Andrade JL, Goncalves LL, Strunz C, Ramos DS, Polli D, Pugliese V, Rodrigues AC, Furtado MS, Carrilho FJ, D'Albuquerque LA. Serum B-type natriuretic peptide in the initial workup of patients with new onset ascites: a diagnostic accuracy study. Hepatology. 2014 Mar;59(3):1043-51. doi: 10.1002/hep.26643. Epub 2014 Jan 13. PMID 23907731